CLINICAL TRIAL: NCT03917160
Title: A Randomized Controlled Trial to Evaluate the Effect of Abdominal EMS (Electrical Muscle Stimulation) on AWR (Abdominal Wall Restoration) in Post - Partum Women
Brief Title: Evaluate the Effect of Abdominal Electrical Muscle Stimulation on Abdominal Wall Restoration in Post - Partum Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InMode MD Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DO608427A
Record Dates: First submitted 2019-04-12; First posted 2019-04-16 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-10

CONDITIONS: Abdominal Wall Restoration; Diastasis Recti

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- EMS treatment (Experimental): Subjects will undergo treatment with EMS and measurements
  Interventions: Device: EMS device
- Control (No Intervention): Subjects will undergo measurements only

INTERVENTIONS:
Device: EMS device — EMS treatment will be performed
  Arms: EMS treatment

SUMMARY:
The objective of the study is to evaluate the safety and efficacy of Abdominal EMS (Electrical Muscle Stimulation) on AWR (Abdominal Wall Restoration) in Post - Partum Women

ELIGIBILITY:
Inclusion Criteria:

* - Post-partum women aged 18-45 years with symptoms of diastasis recti and weakness of the linea alba
* Informed Consent Form signed by the subject.
* BMI interval: 18.5 ≤ BMI ≤ 32 (normal to overweight, but not obese).
* Willing to follow the treatment and follow-up schedule and post-treatment care instructions.
* Willing to have photographs and images taken of the treated areas to be used de-identified in evaluations, publications and presentations.
* In addition, negative urine pregnancy test as tested before each treatment and at the last visit for women with childbearing potential (e.g. not menopause).

Exclusion Criteria:

* - Unable to commit to future appointments
* Planning on moving away from the local area within 6 months
* History of other energy-based therapy within one year
* Diffuse pain syndrome or chronic pain requiring daily narcotics
* Active electrical implant/device in any region of the body, including pacemaker or internal defibrillator
* Permanent implant in the treated area such as metal plates, screws or silicon, metal piercing or other.
* Current or history of skin cancer, or current condition of any other type of cancer, or pre-malignant moles.
* Severe concurrent conditions, such as cardiac disorders, sensory disturbances, epilepsy, uncontrolled hypertension, and liver or kidney diseases.
* History of skin disorders, keloids, abnormal wound healing, as well as very dry and fragile skin.
* History of bleeding coagulopathies or use of anticoagulants except for low-dose aspirin.
* Patients with history of diseases stimulated by heat, such as recurrent Herpes Simplex in the treatment area, may be treated only following a prophylactic regimen.
* Impaired immune system due to immunosuppressive diseases such as AIDS and HIV or use of immunosuppressive medications.
* Pregnancy.
* Poorly controlled endocrine disorders, such as Diabetes, or thyroid dysfunction and hormonal virilization.
* Isotretinoin (Accutane) within last 6 months.
* Any active condition in the treatment area, such as sores, Psoriasis, eczema, and rash, open lacerations, abrasions or lesions, infection in the area to be treated, current urinary tract infection or pelvic infection, uterine prolapse, cystocele, rectocele.
* Any surgical procedure in the treatment area within the last 12 months or before complete healing.
* Having received treatment with light, laser, RF, or other devices in the treated area within 2-3 weeks for non-ablative procedures, and 6-12 weeks for ablative fractional laser resurfacing (according to treatment severity) prior to treatment, except special recommendations.
* Use of non-steroidal anti-inflammatory drugs (NSAIDS, e.g., ibuprofen-containing agents) one week before and after each treatment session, as per the practitioner's discretion.
* As per the practitioner's discretion, refrain from treating any condition which might make it unsafe for the patient.
* Any therapies or medications which may interfere with the use of the study device.
* Compromised health as determined by the study doctor.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Postpartum women
Enrollment: 60 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Change in inter-recti distance (IRD), measured via Magnetic Resonance Imaging. | 1 month
  Up to 5 subjects will undergo MRI to evaluate effect of the treatment
Change in inter-recti distance (IRD), measured via UltraSound Imaging to evaluate effect of the treatment | 1 Month, 3 Months, 6 Months

SECONDARY OUTCOMES:
Change in Urogynecological Complaints measured using the Pelvic Floor Distress Inventory. | 1 Month, 3 Months, 6 Months
  Pelvic Floor Distress Inventory - The PFDI-20 is both a symptom inventory and a measure of the degree of bother and distress (quality-of-life) caused by pelvic floor symptoms.
Change in Severity of Lumbopelvic and/or Abdominal Pain measured by Visual Analog Scale. | 1 Month, 3 Months, 6 Months
  Pain will be assessed based on the Numerical Scale Response (NSR).
Investigator satisfaction | 1 Month, 3 Months, 6 Months
  Satisfaction assessment will be performed by the study investigator using using 0 - 4 -points Likert scale
Subject improvement and satisfaction | 1 Month, 3 Months, 6 Months
  Improvement and satisfaction assessment will be performed independently by the subject using 0 - 4 -points Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Henri Ramirez, MD, Principal Investigator — Southern Oklahoma Women's Health 731 12th Ave NW Suite 201 Ardmore, OK 73401
Locations (2):
- United States (2):
  - Southern Oklahoma Women's Health, Ardmore, Oklahoma
  - Advanced Women's Care of the Lowcountry, PC, Bluffton, South Carolina